CLINICAL TRIAL: NCT06184789
Title: Multiparametric Protocol for Assessment of Intraprocedural Result of MITRACLIP Procedure
Acronym: IPCLIP-2020
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Agricola Eustachio, Principal Investigator, IRCCS San Raffaele
Other Study IDs: INTRAPROCEDURAL-CLIP-2020
Record Dates: First submitted 2023-12-15; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Residual Mitral Regurgitation
Keywords: MitraClip; Residual Mitral Regurgitation; Mitral Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Echocardiographic assessment — Echocardiographic and hemodynamics assessment of Mitraclip results

SUMMARY:
Quantification of residual mitral regurgitation (MR) after MitraClip may be challenging. Quantitative methods for severity assessment may be inaccurate and recent recommendations suggest an assessment of changes in both hemodynamic and echocardiographic parameters, but an established prospectively validated approach is still lacking.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either degenerative or functional, severe or moderate to severe mitral regurgitation (MR) undergoing percutaneous edge-to-edge repair at San Raffaele Hospital from April 2019.

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with either degenerative or functional, severe or moderate to severe mitral regurgitation (MR) undergoing percutaneous edge-to-edge repair at San Raffaele Hospital from April 2019.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of multiparametric assessment of mitral regurgitation ofter Mitraclip | one month

CONTACTS AND LOCATIONS:
Locations (1):
- IRCSS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided